CLINICAL TRIAL: NCT02821533
Title: Chemoembolization for Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor case accrual
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon Yu, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIR-13-04
Record Dates: First submitted 2016-06-07; First posted 2016-07-01 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Cisplatin; Antineoplastic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TACE using a high dose of cisplatin (Other): Two consecutive treatments at two months apart will be given. A delay in the second treatment is allowed if patients do not recover to an acceptable state for subsequent cycle of treatment. Two treatment sessions at one month apart may be required for each complete treatment to cover all lesions when the lesions are diffusely distributed and involving both lobes.
  Interventions: Procedure: TACE; Drug: Cisplatin

INTERVENTIONS:
Procedure: TACE — TACE is performed under local anesthesia with right femoral puncture. The feeding lobar hepatic artery is selectively catheterized for drug delivery.
Drug: Cisplatin — Cisplatin will be mixed with a mixture of Lipiodol and ethanol (LEM), which consists of 33% ethanol by volume in Lipiodol, in a ratio of 2mg cisplatin per mL of LEM, and delivered through catheters or microcatheters to the tumors until there is flow reduction at the tumor feeders. The total dose of cisplatin given in each treatment session is limited to 100mg (50mL LEM) in each treatment session. The usual volume of LEM delivered will be 20 - 30 mL.
  Other Names: chemotherapeutic agent

SUMMARY:
The aim of the current study is to study the safety and effectiveness of TACE using a high dose of cisplatin for treatment of HCC. It is hypothesized that the formulation is safe and it improves the therapeutic effect of conventional TACE.

DETAILED DESCRIPTION:
Most patients with HCC are diagnosed at an intermediate and advanced stage when the tumors become unresectable, transcatheter arterial chemoembolisation (TACE) has been widely accepted as a standard treatment for them in most international management protocols. The therapeutic effect of TACE in terms of objective tumor response is variable and modest (27%-40%), indicating that there is actually much room for improvement in the treatment. Internationally, high doses and combination of chemotherapeutic agents are being routinely and widely used for TACE in major medical centers. Locally, a low dose of cisplatin (10mg) has been used as the chemotherapeutic agent for TACE in Hong Kong. There is evidence showing that the component of chemotherapeutic agent in TACE does play a significant role in the treatment effect of TACE. In an attempt to improve the treatment effect of TACE, the investigators propose a formulation of TACE using a high dose of cisplatin as chemotherapeutic agent.

ELIGIBILITY:
Inclusion Criteria:

Patient factor

1. Age > 18
2. Child-Pugh A or B cirrhosis
3. ECOG performance status Grade 2 or below
4. No serious concurrent medical illness
5. No prior treatment for HCC except for liver resection
6. Creatinine clearance >55ml/min.

Tumor factor

1. HCC diagnosed by typical enhancement patterns on cross sectional imaging or histology.
2. Unresectable and locally advanced disease without extra-hepatic disease
3. Massive expansive tumor type with measurable lesion on CT
4. Total tumor mass < 50% liver volume
5. Largest tumor of greatest dimension ≤ 15cm

Exclusion Criteria:

Patient factor

1. Serum creatinine level > 130 umol/L
2. Presence of biliary obstruction not amenable to percutaneous drainage
3. Child-Pugh C cirrhosis

Evidence of impaired liver function

1. History of hepatic encephalopathy, or
2. Intractable ascites not controllable by medical therapy, or
3. History of variceal bleeding within last 3 months, or
4. Serum total bilirubin level > 40 umol/L, or
5. Serum albumin level < 30g/L, or
6. INR > 1.3

Tumor factor

1. Presence of extrahepatic metastasis
2. Infiltrative lesion
3. Diffuse lesion

Vascular complications

1. Hepatic artery thrombosis, or
2. Partial or complete thrombosis of the main portal vein, or
3. Tumor invasion of portal branch of contralateral lobe, or
4. Hepatic vein tumor thrombus, or
5. Significant arterioportal shunt, or
6. Significant arteriovenous shunt

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-02; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Tumor response | 3 months after treatment
  CT scan abdomen will be performed 3 months after the first treatment. Tumor response by CT was classified into complete response (CR), partial response (PR), static disease (SD, and progressive disease (PD) according to European Association for the Study of the Liver (EASL) necrosis guidelines,

SECONDARY OUTCOMES:
overall survival | 30 days after treatment
  No further treatment was given when there was deterioration in liver function or performance status meeting the exclusion criteria

CONTACTS AND LOCATIONS:
Overall Officials: Simon Yu, Principal Investigator — DIIR, CUHK, Hong Kong
Locations (1):
- Department of Imaging and Interventional Radiology, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No